CLINICAL TRIAL: NCT01466933
Title: Design, Implementation and Evaluation of a Parent Support/Counselling Program With a Focus on Responsive Stimulation for Infants and Young Children in Rural Bangladesh
Brief Title: Responsive Parenting Program for Infants in Rural Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Save the Children (Other)
Responsible Party: Principal Investigator, Frances Aboud, Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB#420-0510
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Child Development
Keywords: parenting intervention; child development; low and middle income countries
MeSH Terms: interventions — Child Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Community-based (Experimental): Community trained peer educator delivers parenting sessions to mothers in the village on a monthly basis
  Interventions: Behavioral: Responsive parenting
- Government-based (Active Comparator): Government community health workers, trained, deliver the intervention to mothers in the village
  Interventions: Behavioral: Child Development
- Control (No Intervention): Mothers receive the standard care which is a visit from the health worker

INTERVENTIONS:
Behavioral: Responsive parenting — On a monthly basis, mothers meet with the peer educator to learn about ways to provide a hygienic environment (hand-washing), proper diverse diet (family foods, breast milk), play materials and conversation to stimulation their child's cognitive and language development. Mothers practice with their child and are coached by the peer educator.
  Arms: Community-based
Behavioral: Child Development — On a monthly basis, mothers meet with the government worker to learn about ways to provide a hygienic environment (hand-washing), proper diverse diet (family foods, breast milk), play materials and conversation to stimulation their child's cognitive and language development.
  Arms: Government-based

SUMMARY:
Children of mothers in the intervention parenting program are expected to show benefits over the standard care control group in terms of better cognitive/language development, less recent illness, and better height for age. The mothers assigned to the intervention parenting program are expected to evidence higher levels of home stimulation, better health prevention, and better dietary diversity, along with more accurate knowledge of child development.

DETAILED DESCRIPTION:
There are actually two intervention groups: in one the program is delivered by trained peer educators from the village, and in the other the program is delivered by trained government personnel.

ELIGIBILITY:
Inclusion Criteria:

* mother has a child 6 to 14 months of age
* mother willing to learn about child care

Exclusion Criteria:

* not severely disabled

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 474 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Bayley scales of infant development | 12 months
  Cognitive, receptive language and expressive language items will be administered to the child and scored as pass/fail with a total score calculated for each subtest and the total.

SECONDARY OUTCOMES:
HOME Inventory | 12 months
  45 items assessing through observation and interview opportunities for stimulation in the home.
Mother-Child picture talk | 12 months
  Mothers' responsive talk while looking at pictures with her child.
Dietary diversity | 12 months
  Number out of 7 categories of food, based on Mothers recall foods fed to their child over a 24-hour period.
Child development knowledge of mother | 12 months
  Mothers report the age when they expect children to start acquiring 10 psychosocial skills, e.g. recognize its mother.
height for age | 12 months
  height for age z score is derived from the current WHO growth standards

CONTACTS AND LOCATIONS:
Overall Officials: Frances Aboud, PhD, Principal Investigator — McGill University
Locations (1):
- Save the Children district office, Kushtia, Bangladesh